CLINICAL TRIAL: NCT05751200
Title: Safety and Efficacy of Aortic Root Reinforcement Combined With Vascular Grafts Eversion and built-in Procedure (XJ-procedure) in Patients With Acute Type A Aortic Dissection (ADVANCED-XJ ): an Investigator-initiated, Single-center, Cohort Study
Brief Title: Safety and Efficacy of Aortic Root Reinforcement Combined With Vascular Grafts Eversion and built-in Procedure (XJ-procedure) in Patients With Acute Type A Aortic Dissection (ADVANCED-XJ )
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-150
Record Dates: First submitted 2023-02-14; First posted 2023-03-02 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Type A Aortic Dissection
Keywords: Type A Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CARS group: In the CARS group, 3-0 polypropylene was used to suture the proximal end of aortic with the vascular grafts continuously, followed by one interrupted suture loop of 3-0 polypropylene for reinforcement.
  Interventions: Other: No Intervention.
- XJ-procedure group: In the XJ-procedure group, a 1.5-2cm wide bovine pericardial patch and graft ring were placed inside and outside the aortic root and against the aortic wall, respectively, and continuously sutured near the commissure using 5-0 polypropylene. Then an eversion about 15mm of vascular graft was intermittently sutured to full layers of aortic vascular with 2-0 pad polyester sutures. Finally, the eversion and aortic wall were continuously sutured together in one more turn.
  Interventions: Other: No Intervention.

INTERVENTIONS:
Other: No Intervention. — No Intervention.

SUMMARY:
This is a retrospective study based on the data available in our hospital database for ATAAD patients from January 2020 to December 2021. These patients were divided into two groups according to the surgical procedures of aortic root. This study compared baseline data, perioperative and short-term follow-up results between the two groups to evaluate the efficacy and safety of XJ-procedure in ATAAD.

DETAILED DESCRIPTION:
Acute type A aortic dissection (ATAAD) is a life-threatening disease with high mortality. Surgery remains the gold standard for the treatment of ATAAD. In recent years, ATAAD is still a persistent challenge for cardiovascular surgeons. This is a retrospective study based on the data available in our hospital database for ATAAD patients undergoing total aortic arch replacement with elephant trunk stent under cryogenic stop circulation from January 2020 to December 2021. These patients were divided into two groups according to the surgical procedures of aortic root: continuous aortic root suture group (CARS group); "aortic root reinforcement combined with vascular grafts eversion and built-in", which was created by our group and to be named as XJ-procedure (XJ-procedure group, XJ is an acronym for Xi'an Jiaotong University). The main outcome was defined as 30-day mortality. Secondary outcomes included the postoperative bleeding necessitating re-operation and the incidence of anastomotic pseudoaneurysm, residual aortic root dissection and severe aortic regurgitation before discharge and at 3 and 6 months after the operation. This study compared baseline data, perioperative and short-term follow-up results between the two groups to evaluate the efficacy and safety of XJ-procedure in ATAAD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ATAAD by computed tomography angiography (CTA) from January 2020 to December 2021 in the First Affiliated Hospital of Xi'an Jiaotong University
* Mild to moderate aortic root involvement
* Aortic arch involvement undergoing Sun's procedure

Exclusion Criteria:

* Patients with severe aortic root involvement (root diameter >45 mm, root tear, severe disruption of aortic root, concomitant valve disease)
* The Bentall, Wheat or David procedure performed
* Recurrent ATAAD
* Preoperative severe brain complications (cerebral infarction, cerebral hemorrhage, coma, etc.)
* Mal-perfusion of abdominal organs or lower extremities >12 h
* Incomplete clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolled patients who were diagnosed with ATAAD by computed tomography angiography (CTA) from January 2020 to December 2021 in the First Affiliated Hospital of Xi'an Jiaotong University. Inclusion criteria included mild to moderate aortic root involvement, combined with aortic arch involvement undergoing Sun's procedure. The exclusion criteria included severe aortic root involvement (root diameter >45 mm, root tear, severe disruption of aortic root, concomitant valve disease); the Bentall, Wheat or David procedure performed; recurrent ATAAD; preoperative severe brain complications (cerebral infarction, cerebral hemorrhage, coma, etc.), mal-perfusion of abdominal organs or lower extremities >12 h and incomplete clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
30-day mortality | Within 30 days after the surgery
  Patients died within 30 days after the surgery. Data were obtained from the medical records.

SECONDARY OUTCOMES:
The postoperative bleeding necessitating re-operation | About 2 weeks after the surgery.
  Postoperative bleeding necessitated reoperation during hospitalization. Data were obtained from the surgical records and medical records.
Change in the incidence of anastomotic pseudoaneurysm | About 2 weeks after surgery, 3-month and 6-month follow-up.
  The occurrence of anastomotic pseudoaneurysm was examined by postoperative computed tomography angiography examination.
Change in the incidence of residual aortic root dissection | About 2 weeks after surgery, 3-month and 6-month follow-up.
  The occurrence of residual aortic dissection was examined by postoperative computed tomography angiography examination.
Change in the incidence of severe aortic regurgitation | About 2 weeks after surgery, 3-month and 6-month follow-up.
  The occurrence of aortic valve regurgitation greater than grade2+, which was decided by cardiac ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Zhao C, Li B, Yan P, Zhang Y, Li Y, Wang Q, He X, Zheng X, Yan Y. Aortic Root Reinforcement Combined with Vascular Grafts Eversion and Built-in Procedure (XJ-Procedure) for Acute Type A Aortic Dissection Surgery. Adv Ther. 2023 Dec;40(12):5354-5365. doi: 10.1007/s12325-023-02655-2. Epub 2023 Oct 4. PMID 37789228